CLINICAL TRIAL: NCT05546476
Title: A PHASE 2, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO INVESTIGATE THE EFFICACY, SAFETY AND TOLERABILITY OF PONSEGROMAB IN PATIENTS WITH CANCER, CACHEXIA, AND ELEVATED CONCENTRATIONS OF GDF-15, FOLLOWED BY AN OPTIONAL OPEN-LABEL TREATMENT PERIOD (PROACC -1)
Brief Title: Study of the Efficacy and Safety of Ponsegromab in Patients With Cancer, Cachexia and Elevated GDF-15
Acronym: PROACC-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C3651003; 2023-510446-24-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-08-12; First posted 2022-09-19 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer; Pancreatic Cancer; Colorectal Cancer; Loss of Appetite; Fatigue; Cachexia
Keywords: cancer; anorexia; cachexia; weight loss; loss of appetite; fatigue
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Colorectal Neoplasms; Anorexia; Fatigue; Cachexia; Neoplasms; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind for 12-week double-blind treatment period followed by an up to 1 year optional open-label treatment period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Double-Blind ponsegromab Treatment low dose followed by Open Label ponsegromab Treatment (Experimental): ponsegromab low dose subcutaneous injection every 4 weeks
  Interventions: Drug: ponsegromab
- Double-Blind Placebo Treatment followed by Open-Label ponsegromab Treatment (Placebo Comparator): Match placebo subcutaneous injection every 4 weeks
  Interventions: Drug: Placebo for ponsegromab
- Double-Blind ponsegromab Treatment medium dose followed by Open Label ponsegromab Treatment (Experimental): ponsegromab medium dose subcutaneous injection every 4 weeks
  Interventions: Drug: ponsegromab
- Double-Blind ponsegromab Treatment high dose followed by Open Label ponsegromab Treatment (Experimental): ponsegromab high dose subcutaneous injection every 4 weeks
  Interventions: Drug: ponsegromab

INTERVENTIONS:
Drug: ponsegromab — Double-Blind ponsegromab Treatment followed by Open Label ponsegromab Treatment
  Arms: Double-Blind ponsegromab Treatment high dose followed by Open Label ponsegromab Treatment; Double-Blind ponsegromab Treatment low dose followed by Open Label ponsegromab Treatment; Double-Blind ponsegromab Treatment medium dose followed by Open Label ponsegromab Treatment
Drug: Placebo for ponsegromab — Double-Blind placebo Treatment followed by Open Label ponsegromab Treatment
  Arms: Double-Blind Placebo Treatment followed by Open-Label ponsegromab Treatment

SUMMARY:
Study to evaluate the efficacy, safety and tolerability of ponsegromab compared to placebo in patients with cancer, cachexia, and elevated GDF 15.

DETAILED DESCRIPTION:
A 12 week double blind study to evaluate the efficacy, safety and tolerability of ponsegromab compared to placebo in patients with cancer, cachexia, and elevated GDF 15.

During the initial 12-week treatment period (Part A), a total of 3 doses of ponsegromab or placebo will be administered 4 weeks apart subcutaneously. Each dose contains two injections. Part B is an optional open-label treatment period consisting of ponsegromab administered every 4 weeks subcutaneously for up to one year. Part B does not include placebo.

Assessments include:

* Body weight measurements
* Measure the impact of ponsegromab compared to placebo on physical activity.
* Measure the impact of ponsegromab compared to placebo on appetite, fatigue, nausea, vomiting and physical function questionnaires.
* Blood samples to evaluate safety and additional endpoints including the amount of study drug in the blood and the effects of the study drug on levels of GDF15
* Up to 3 additional blood samples (two samples during Part A and one sample during Part B, if relevant) in a subset of participants as part of a substudy for more comprehensive assessment of the amount of study drug in the blood and of the effects of the study drug on levels of GDF-15.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented active diagnosis of non-small cell lung, pancreatic, colorectal cancer
* Cachexia defined by Fearon criteria of weight loss
* Serum GDF-15 concentrations
* Signed informed consent
* ECOG PS ≤3 with life expectancy of at least 4 months to be able to complete Part A.

Key Exclusion Criteria:

* Receiving tube feedings or parenteral nutrition at the time of Screening or Randomization.
* Current active reversible causes of decreased food intake.
* Cachexia caused by other reasons.
* History of allergic or anaphylactic reaction to any therapeutic or diagnostic monoclonal antibody.
* inadequate liver function
* renal disease requiring dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2025-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (78):
- United States (19):
  - CARTI Conway, Conway, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - CARTI North Little Rock, North Little Rock, Arkansas
  - CARTI Stuttgart, Stuttgart, Arkansas
  - Pacific Cancer Medical Center INC, Anaheim, California
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Emad Ibrahim,MD,INC., Redlands, California
  - Providence Medical Foundation, Santa Rosa, California
  - IU Health Arnett Cancer Center, Lafayette, Indiana
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Oregon Health and Science University: Center for Health and Healing 1, Portland, Oregon
  - Oregon Health and Science University: Center for Health and Healing 2, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Carta - Clinical Associates in Research Therapeutics of America, LLC, San Antonio, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Wenatchee Valley Hospital, Wenatchee, Washington
- Australia (4):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Orange Hospital, Orange, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Western Health-Sunshine & Footscray Hospitals, St Albans, Victoria
- Bulgaria (8):
  - Complex Oncology Center - Burgas, Burgas
  - Specialized Hospital for Active Treatment of Oncology - Haskovo, Haskovo
  - Complex Oncology Center - Ruse EOOD, Rousse
  - Complex Oncology Center - Shumen, Shumen
  - Multiprofile Hospital for Active Treatment Serdika EOOD, Sofia
  - MHAT for Women's Health Nadezhda, Sofia
  - University Multiprofile Hospital for Active Treatment Sofiamed, Sofia
  - Complex Oncology Center - Vratsa, Vratsa
- Canada (4):
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CIUSSS- saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Centre intégré de santé et de services sociaux du Bas Saint-Laurent- Hôpital régional de Rimouski, Rimouski, Quebec
- China (10):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The 2nd Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Hungary (4):
  - Bacs-Kiskun Varmegyei Oktatokorhaz, Kecskemét, Bács-Kiskun county
  - Jász-Nagykun-Szolnok Vármegyei Hetényi Géza Kórház, Szolnok, Jász-Nagykun-Szolnok
  - Semmelweis Egyetem, Budapest
  - Országos Korányi Pulmonológiai Intézet, Budapest
- Japan (8):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Kanagawa cancer center, Yokohama, Kanagawa
  - Aichi Cancer Center Hospital, Nagoya, Nagoya, Aichi
  - Shizuoka Cancer Center, Nagaizumi-cho, Shizuoka
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto
  - The Cancer Institute Hospital of JFCR, Tokyo
- Poland (4):
  - Centrum Badań Klinicznych Jagiellońskie Centrum Innowacji sp. z o.o., Krakow, Lesser Poland Voivodeship
  - Regionalny Szpital Specjalistyczny im. Dr. Wladyslawa Bieganskiego, Grudziądz
  - NZOZ "Vegamed", Katowice
  - Specjalistyczna Praktyka Lekarska Slawomir Mandziuk, Lublin
- Slovakia (6):
  - Fakultna nemocnica s poliklinikou F. D. Roosevelta Banska Bystrica, Banská Bystrica
  - Univerzitna nemocnica Bratislava, Nemocnica Ruzinov, Bratislava
  - Narodny onkologicky ustav, II. Onkologicka klinika LFUK a NOU, Bratislava
  - Fakultna nemocnica s poliklinikou Nove Zamky, Nové Zámky
  - Nemocnica na okraji mesta, n.o., Partizánske
  - Fakultna nemocnica Trnava, Trnava
- Spain (6):
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès, Barcelona [barcelona]
  - Institut Català d'Oncologia - L'Hospitalet, L'Hospitalet de Llobregat, Catalunya [cataluña]
  - Hospital Son Llàtzer, Palma, Illes Balears [islas Baleares]
  - Fundación Instituto Valenciano de Oncología, Valencia, Valenciana, Comunitat
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (5):
  - Chi Mei Hospital - Liouying Branch, Tainan, Tainan
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Groarke JD, Crawford J, Collins SM, Lubaczewski S, Roeland EJ, Naito T, Hendifar AE, Fallon M, Takayama K, Asmis T, Dunne RF, Karahanoglu I, Northcott CA, Harrington MA, Rossulek M, Qiu R, Saxena AR. Ponsegromab for the Treatment of Cancer Cachexia. N Engl J Med. 2024 Dec 19;391(24):2291-2303. doi: 10.1056/NEJMoa2409515. Epub 2024 Sep 14. PMID 39282907
- [Derived] Groarke JD, Crawford J, Collins SM, Lubaczewski SL, Breen DM, Harrington MA, Jacobs I, Qiu R, Revkin J, Rossulek MI, Saxena AR. Phase 2 study of the efficacy and safety of ponsegromab in patients with cancer cachexia: PROACC-1 study design. J Cachexia Sarcopenia Muscle. 2024 Jun;15(3):1054-1061. doi: 10.1002/jcsm.13435. Epub 2024 Mar 18. PMID 38500292
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3651003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 187 participants were enrolled in this study. This study had 2 parts: Part A and Part B. On completion of Part A, participants had the opportunity to enter open-label extension period Part B (optional). Results are reported on the primary completion date of the study. At this milestone Part A analysis (primary and secondary outcome measures) was final.
Groups:
- Part A: Placebo/ Part B: Ponsegromab 400 mg: Part A: Participants were randomized to receive placebo matching to Ponsegromab subcutaneously (SC) once in every 4 weeks (Q4W) up to 12 weeks (total of 3 doses). Part B: On completion of Part A, participants had the opportunity to receive open label Ponsegromab 400 mg Q4W SC for up to 1 year.
- Part A: Ponsegromab 100 mg/ Part B: Ponsegromab 400 mg: Part A: Participants were randomized to receive Ponsegromab 100 milligrams (mg) SC Q4W up to 12 weeks (total of 3 doses). Part B: On completion of Part A, participants had the opportunity to receive open label Ponsegromab 400 mg Q4W SC for up to 1 year.
- Part A: Ponsegromab 200 mg/ Part B: Ponsegromab 400 mg: Part A: Participants were randomized to receive Ponsegromab 200 mg SC Q4W up to 12 weeks (total of 3 doses). Part B: On completion of Part A, participants had the opportunity to receive open label Ponsegromab 400 mg Q4W SC for up to 1 year.
- Part A: Ponsegromab 400 mg/ Part B: Ponsegromab 400 mg: Part A: Participants were randomized to receive Ponsegromab 400 mg SC Q4W up to 12 weeks (total of 3 doses). Part B: On completion of Part A, participants had the opportunity to receive open label Ponsegromab 400 mg Q4W SC for up to 1 year.
Period: Period 1: Part A
Arm/Group | Part A: Placebo/ Part B: Ponsegromab 400 mg | Part A: Ponsegromab 100 mg/ Part B: Ponsegromab 400 mg | Part A: Ponsegromab 200 mg/ Part B: Ponsegromab 400 mg | Part A: Ponsegromab 400 mg/ Part B: Ponsegromab 400 mg
Started | 45 | 46 | 46 | 50
Completed | 32 | 32 | 39 | 34
Not Completed | 13 | 14 | 7 | 16
Not completed — Adverse Event | 2 | 0 | 0 | 1
Not completed — Death | 4 | 4 | 5 | 6
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Progressive disease | 3 | 5 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 2
Not completed — Global deterioration of health status | 2 | 2 | 1 | 4
Not completed — Other: Unspecified | 0 | 2 | 0 | 0
Period: Period 2: Part B
Arm/Group | Part A: Placebo/ Part B: Ponsegromab 400 mg | Part A: Ponsegromab 100 mg/ Part B: Ponsegromab 400 mg | Part A: Ponsegromab 200 mg/ Part B: Ponsegromab 400 mg | Part A: Ponsegromab 400 mg/ Part B: Ponsegromab 400 mg
Started | 26 | 27 | 35 | 29
Completed | 0 | 0 | 0 | 0
Not Completed | 26 | 27 | 35 | 29
Not completed — Ongoing | 26 | 27 | 35 | 29

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received.
Groups:
- Part A: Placebo/ Part B: Ponsegromab 400 mg: Part A: Participants were randomized to receive placebo matching to Ponsegromab SC Q4W up to 12 weeks (total of 3 doses). Part B: On completion of Part A, participants had the opportunity to receive open label Ponsegromab 400 mg Q4W SC for up to 1 year.
- Part A: Ponsegromab 100 mg/ Part B: Ponsegromab 400 mg: Part A: Participants were randomized to receive Ponsegromab 100 mg SC Q4W up to 12 weeks (total of 3 doses). Part B: On completion of Part A, participants had the opportunity to receive open label Ponsegromab 400 mg Q4W SC for up to 1 year.
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo/ Part B: Ponsegromab 400 mg | Part A: Ponsegromab 100 mg/ Part B: Ponsegromab 400 mg | Part A: Ponsegromab 200 mg/ Part B: Ponsegromab 400 mg | Part A: Ponsegromab 400 mg/ Part B: Ponsegromab 400 mg | Total
Number analyzed (Participants) | 45 | 46 | 46 | 50 | 187
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (11.26) | 70.1 (9.38) | 65.9 (9.61) | 66.1 (9.93) | 66.4 (10.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 15 | 18 | 69
  Male | 28 | 27 | 31 | 32 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 5 | 9
  Not Hispanic or Latino | 43 | 42 | 44 | 43 | 172
  Unknown or Not Reported | 1 | 3 | 0 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 18 | 19 | 18 | 15 | 70
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 26 | 27 | 28 | 35 | 116
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part A: Change From Baseline in Body Weight at Week 12
Description: Body weight was measured in kilograms using a calibrated weighing scale. Baseline was defined as the last average of the duplicate measurements prior to, or on Day 1. The average of the duplicate body weights collected at assessment time was considered. The posterior medians and 90 percent (%) credible intervals (5th and 95th percentiles of the relevant posterior distribution) were reported for each randomized dose (including placebo). 4-Parameter maximal effect (E max) model: change from baseline = E 0 + (E max * dose^Hill) / (ED 50^Hill + dose^Hill), where E0 is the placebo effect, E max is the maximum effect, ED 50 is the dose producing 50% of the maximum effect, and Hill is the slope parameter. Model utilized a Bayesian methodology with a robustified, informative meta-analytic predictive prior for the placebo change from baseline at week 12.
Time Frame: Baseline, Week 12
Population: Censored analysis set included all evaluable participants. For participants who discontinued study intervention, or received a prohibited procedure or prohibited medication, all observations post-discontinuation, or post-procedure, were censored and treated as missing data. For participants who missed a dose, or received an incomplete dose, all observations post-missed/incomplete dose were censored and treated as missing data.
Measure: Median (90% Confidence Interval); unit: Kilogram
Groups:
- Part A: Placebo: Part A: Participants were randomized to receive placebo matching to Ponsegromab SC Q4W up to 12 weeks (total of 3 doses).
- Part A: Ponsegromab 100 mg: Part A: Participants were randomized to receive Ponsegromab 100 mg SC Q4W up to 12 weeks (total of 3 doses).
- Part A: Ponsegromab 200 mg: Part A: Participants were randomized to receive Ponsegromab 200 mg SC Q4W up to 12 weeks (total of 3 doses).
- Part A: Ponsegromab 400 mg: Part A: Participants were randomized to receive Ponsegromab 400 mg SC Q4W up to 12 weeks (total of 3 doses).
Arm/Group | Part A: Placebo | Part A: Ponsegromab 100 mg | Part A: Ponsegromab 200 mg | Part A: Ponsegromab 400 mg
Number analyzed (Participants) | 45 | 46 | 46 | 50
Kilogram | NA [NA to NA] — Measure Type = Posterior Median = -0.60 Measure of Dispersion = 90% Credible Interval = -1.50 to 0.24 | NA [NA to NA] — Measure Type = Posterior Median = 0.75 Measure of Dispersion = 90% Credible Interval = 0.06 to 1.44 | NA [NA to NA] — Measure Type = Posterior Median = 1.48 Measure of Dispersion = 90% Credible Interval = 0.87 to 2.08 | NA [NA to NA] — Measure Type = Posterior Median = 2.39 Measure of Dispersion = 90% Credible Interval = 1.49 to 3.34
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Ponsegromab 100 mg; Bayesian Emax model was used for statistical calculation. The posterior medians and 90% credible intervals (5th and 95th percentiles of the relevant posterior distribution) were reported for differences relative to placebo). No adjustments were made for multiplicity; Test type: Superiority; Difference in Posterior Median = 1.33, 90% CI 2-sided [0.49 to 2.34]
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: Ponsegromab 200 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in Posterior Median = 2.08, 90% CI 2-sided [1.08 to 3.15]
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: Ponsegromab 400 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in Posterior Median = 3, 90% CI 2-sided [1.68 to 4.34]

2. Secondary Outcome: Part A: Change From Baseline in Physical Activity at Week 12
Description: Physical activity was monitored using accelerometry (wearable digital sensors). Physical activity was categorized as: sedentary activity, non-sedentary physical activity, and moderate to vigorous physical activity. In this outcome measure time for each type of physical activity per day was considered. Baseline was defined as the mean taken over the 8 days of wear during screening. Mean taken over the 8 days of wear before Week 12 was considered. Analysis was performed using mixed models repeated measures (MMRM) model.
Time Frame: Baseline, Week 12
Population: Censored analysis set:all evaluable participants.For participants who discontinued study intervention/received prohibited procedure/ prohibited medication,all observations post-discontinuation/post-procedure,were censored and treated as missing data.For participants who missed dose/received incomplete dose,all observations post-missed/incomplete dose were censored and treated as missing data.''Overall Number of Participants Analyzed'' =participants evaluable for this outcome measure at Week 12.
Measure: Least Squares Mean (90% Confidence Interval); unit: Minutes per day
Arm/Group | Part A: Placebo | Part A: Ponsegromab 100 mg | Part A: Ponsegromab 200 mg | Part A: Ponsegromab 400 mg
Number analyzed (Participants) | 12 | 17 | 16 | 13
Minutes per day
  Time for Sedentary Activity | -1.42 [-72.77 to 69.92] | 51.93 [-9.88 to 113.75] | -39.33 [-101.94 to 23.29] | -3.37 [-72.89 to 66.14]
  Time for Non-Sedentary Physical Activity | -37.73 [-66.14 to -9.32] | 0.03 [-24.88 to 24.95] | -42.09 [-67.63 to -16.56] | 12.11 [-14.87 to 39.10]
  Time for Moderate to Vigorous Physical Activity | -4.45 [-13.91 to 5.02] | 4.07 [-4.18 to 12.32] | 0.05 [-8.29 to 8.39] | 3.67 [-5.37 to 12.71]
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Ponsegromab 100 mg; Sedentary Activity Time: MMRM model included participant as a random term, and baseline, time (as a factor), baseline-by-time interaction, treatment and treatment-by-time interaction, type of therapy [platinum or not at randomization +/- 28 days], and type of cancer as fixed terms, with an unstructured covariance matrix and Kenwood-Roger degrees of freedom; Test type: Superiority; p = 0.8260, MMRM analysis; 1-sided; Difference in LS Mean = 53.36, 90% CI 2-sided [-40.89 to 147.60]
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: Ponsegromab 200 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.2540, MMRM analysis; 1-sided; Difference in LS Mean = -37.9, 90% CI 2-sided [-132.94 to 57.14]
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: Ponsegromab 400 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.4870, MMRM analysis; 1-sided; Difference in LS Mean = -1.95, 90% CI 2-sided [-101.63 to 97.73]
Statistical Analysis 4: Comparison: Part A: Placebo vs Part A: Ponsegromab 100 mg; Non-Sedentary Activity Time: MMRM model included participant as a random term, and baseline, time (as a factor), baseline-by-time interaction, treatment and treatment-by-time interaction, type of therapy [platinum or not at randomization +/- 28 days], and type of cancer as fixed terms, with an unstructured covariance matrix and Kenwood-Roger degrees of freedom; Test type: Superiority; p = 0.0497, MMRM analysis; 1-sided; Difference in LS Mean = 37.76, 90% CI 2-sided [0.07 to 75.46]
Statistical Analysis 5: Comparison: Part A: Placebo vs Part A: Ponsegromab 200 mg; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = 0.5745, MMRM analysis; 1-sided; Difference in LS Mean = -4.36, 90% CI 2-sided [-42.94 to 34.22]
Statistical Analysis 6: Comparison: Part A: Placebo vs Part A: Ponsegromab 400 mg; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = 0.0189, MMRM analysis; 1-sided; Difference in LS Mean = 49.85, 90% CI 2-sided [10.62 to 89.08]
Statistical Analysis 7: Comparison: Part A: Placebo vs Part A: Ponsegromab 100 mg; Moderate to Vigorous Physical Activity Time: MMRM model included participant as a random term, and baseline, time (as a factor), baseline-by-time interaction, treatment and treatment-by-time interaction, type of therapy [platinum or not at randomization +/- 28 days], and type of cancer as fixed terms, with an unstructured covariance matrix and Kenwood-Roger degrees of freedom; Test type: Superiority; p = 0.1302, MMRM analysis; 1-sided; Difference in LS Mean = 8.51, 90% CI 2-sided [-4.00 to 21.03]
Statistical Analysis 8: Comparison: Part A: Placebo vs Part A: Ponsegromab 200 mg; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; p = 0.2780, MMRM analysis; 1-sided; Difference in LS Mean = 4.49, 90% CI 2-sided [-8.18 to 17.16]
Statistical Analysis 9: Comparison: Part A: Placebo vs Part A: Ponsegromab 400 mg; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; p = 0.1529, MMRM analysis; 1-sided; Difference in LS Mean = 8.11, 90% CI 2-sided [-5.01 to 21.23]

3. Secondary Outcome: Part A: Change From Baseline in Mean Activity Level During Maximum 6 Minutes at Week 12
Description: Physical activity was monitored using accelerometry (wearable digital sensors). In this outcome measure mean activity level during maximum 6 minutes was considered. Baseline was defined as the mean taken over the 8 days of wear during screening. Mean taken over the 8 days of wear before Week 12 was considered. Analysis was performed using MMRM model.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (90% Confidence Interval); unit: Arbitrary units per day (au/day)
Arm/Group | Part A: Placebo | Part A: Ponsegromab 100 mg | Part A: Ponsegromab 200 mg | Part A: Ponsegromab 400 mg
Number analyzed (Participants) | 12 | 17 | 16 | 13
Arbitrary units per day (au/day) | 70.81 [-785.82 to 927.45] | -59.46 [-794.41 to 675.49] | 794.96 [39.43 to 1550.48] | 256.43 [-561.29 to 1074.16]
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Ponsegromab 100 mg; MMRM model included participant as a random term, and baseline, time (as a factor), baseline-by-time interaction, treatment and treatment-by-time interaction, type of therapy [platinum or not at randomization +/- 28 days], and type of cancer as fixed terms, with an unstructured covariance matrix and Kenwood-Roger degrees of freedom; Test type: Superiority; p = 0.5762, MMRM analysis; 1-sided; Difference in LS Mean = -130.27, 90% CI 2-sided [-1257.31 to 996.77]
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: Ponsegromab 200 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.1486, MMRM analysis; 1-sided; Difference in LS Mean = 724.14, 90% CI 2-sided [-425.81 to 1874.09]
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: Ponsegromab 400 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.3972, MMRM analysis; 1-sided; Difference in LS Mean = 185.62, 90% CI 2-sided [-997.94 to 1369.18]

4. Secondary Outcome: Part A: Change From Baseline in Total Vector Magnitude at Week 12
Description: Total vector magnitude is a measure of overall physical activity. Baseline was defined as the mean taken over the 8 days of wear during screening. Mean taken over the 8 days of wear before Week 12 was considered. Analysis was performed using MMRM model.
Time Frame: Baseline, Week 12
Population: Censored analysis set: all evaluable participants. For participants who discontinued study intervention/received prohibited procedure/ prohibited medication,all observations post-discontinuation/post-procedure,were censored and treated as missing data.For participants who missed dose/received incomplete dose,all observations post-missed/incomplete dose were censored and treated as missing data.''Overall Number of Participants Analyzed''=participants evaluable for this outcome measure at Week 12
Measure: Least Squares Mean (90% Confidence Interval); unit: Total activity counts/100 per day
Arm/Group | Part A: Placebo | Part A: Ponsegromab 100 mg | Part A: Ponsegromab 200 mg | Part A: Ponsegromab 400 mg
Number analyzed (Participants) | 12 | 17 | 16 | 13
Total activity counts/100 per day | -1919.02 [-3450.37 to -387.68] | -331.76 [-1679.81 to 1016.29] | -2017.57 [-3387.48 to -647.65] | 284.15 [-1175.46 to 1743.77]
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Ponsegromab 100 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0985, MMRM analysis; 1-sided; Difference in LS Mean = 1587.26, 90% CI 2-sided [-443.79 to 3618.31]
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: Ponsegromab 200 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.5315, MMRM analysis; 1-sided; Difference in LS Mean = -98.54, 90% CI 2-sided [-2169.67 to 1972.58]
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: Ponsegromab 400 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0437, MMRM analysis; 1-sided; Difference in LS Mean = 2203.18, 90% CI 2-sided [84.51 to 4321.85]

5. Secondary Outcome: Part A: Change From Baseline in Gait at Week 12
Description: Gait was monitored using accelerometry (wearable digital sensors). Analysis was performed using MMRM model. Gait included: gait speed and 95th percentile of gait speed. Baseline was defined as the mean taken over the 8 days of wear during screening. Mean taken over the 8 days of wear before Week 12 was considered. Analysis was performed using MMRM model.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (90% Confidence Interval); unit: Meter per second (m/s)
Arm/Group | Part A: Placebo | Part A: Ponsegromab 100 mg | Part A: Ponsegromab 200 mg | Part A: Ponsegromab 400 mg
Number analyzed (Participants) | 15 | 19 | 18 | 14
Meter per second (m/s)
  Gait Speed | -0.008 [-0.042 to 0.026] | -0.009 [-0.040 to 0.023] | -0.012 [-0.044 to 0.019] | 0.009 [-0.024 to 0.042]
  95th percentile of gait speed | 0.011 [-0.041 to 0.064] | 0.011 [-0.037 to 0.059] | -0.015 [-0.063 to 0.033] | 0.021 [-0.030 to 0.072]
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Ponsegromab 100 mg; Gait Speed: MMRM model included participant as a random term, and baseline, time (as a factor), baseline-by-time interaction, treatment and treatment-by-time interaction, type of therapy [platinum or not at randomization +/- 28 days], and type of cancer as fixed terms, with an unstructured covariance matrix and Kenwood-Roger degrees of freedom; Test type: Superiority; p = 0.5052, MMRM analysis; 1-sided; Difference in LS Mean = 0, 90% CI 2-sided [-0.046 to 0.045]
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: Ponsegromab 200 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.5599, MMRM analysis; 1-sided; Difference in LS Mean = -0.004, 90% CI 2-sided [-0.050 to 0.042]
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: Ponsegromab 400 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.2770, MMRM analysis; 1-sided; Difference in LS Mean = 0.017, 90% CI 2-sided [-0.030 to 0.064]
Statistical Analysis 4: Comparison: Part A: Placebo vs Part A: Ponsegromab 100 mg; 95th Percentile of Gait Speed: MMRM model included participant as a random term, and baseline, time (as a factor), baseline-by-time interaction, treatment and treatment-by-time interaction, type of therapy [platinum or not at randomization +/- 28 days], and type of cancer as fixed terms, with an unstructured covariance matrix and Kenwood-Roger degrees of freedom; Test type: Superiority; p = 0.5047, MMRM analysis; 1-sided; Difference in LS Mean = 0, 90% CI 2-sided [-0.071 to 0.070]
Statistical Analysis 5: Comparison: Part A: Placebo vs Part A: Ponsegromab 200 mg; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p = 0.7316, MMRM analysis; 1-sided; Difference in LS Mean = -0.026, 90% CI 2-sided [-0.097 to 0.045]
Statistical Analysis 6: Comparison: Part A: Placebo vs Part A: Ponsegromab 400 mg; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p = 0.4145, MMRM analysis; 1-sided; Difference in LS Mean = 0.01, 90% CI 2-sided [-0.063 to 0.082]

6. Secondary Outcome: Part A: Change From Baseline in Functional Assessment of Anorexia-Cachexia Therapy- Anorexia and Cachexia Subscale (FAACT-ACS) at Week 12
Description: FAACT-ACS is a 12-item symptom-specific subscale to measure participants' concerns about their anorexia (appetite) or cachexia (weight) for past 7 days. Each item was scored from 0 to 4, where 0= not at all, 1= a little bit, 2= somewhat, 3= quite a bit, and 4= very much. The total FAACT-ACS score ranged from 0 to 48. Higher scores are associated with a higher health-related quality of life. FAACT-ACS was analyzed using an MMRM model.
Time Frame: Baseline (prior to dose on Day 1), Week 12
Population: as for outcome 2
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Part A: Placebo | Part A: Ponsegromab 100 mg | Part A: Ponsegromab 200 mg | Part A: Ponsegromab 400 mg
Number analyzed (Participants) | 30 | 27 | 33 | 27
Units on a scale | 0.52 [-1.60 to 2.63] | 4.76 [2.54 to 6.97] | 1.15 [-0.90 to 3.20] | 4.63 [2.40 to 6.85]
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Ponsegromab 100 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0114, MMRM analysis; 1-sided; Difference in LS Mean = 4.24, 90% CI 2-sided [1.19 to 7.28]
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: Ponsegromab 200 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.3600, MMRM analysis; 1-sided; Difference in LS Mean = 0.64, 90% CI 2-sided [-2.30 to 3.57]
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: Ponsegromab 400 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0138, MMRM analysis; 1-sided; Difference in LS Mean = 4.11, 90% CI 2-sided [1.06 to 7.17]

7. Secondary Outcome: Part A: Change From Baseline in FAACT- 5-Item Anorexia Symptom Scale (5IASS) at Week 12
Description: FAACT-5IASS is a 5-item subscale to measure participants' perceptions of anorexia (appetite) concerns for past 7 days. Each item was scored from 0 to 4, where 0= not at all, 1= a little bit, 2= somewhat, 3= quite a bit, and 4= very much. The total FAACT-5IASS score ranged from 0 to 20. Higher scores are associated with a higher health-related quality of life. FAACT-5IASS was analyzed using an MMRM model.
Time Frame: Baseline (prior to dose on Day 1), Week 12
Population: as for outcome 2
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Part A: Placebo | Part A: Ponsegromab 100 mg | Part A: Ponsegromab 200 mg | Part A: Ponsegromab 400 mg
Number analyzed (Participants) | 30 | 27 | 33 | 27
Units on a scale | 0.15 [-0.97 to 1.27] | 2.50 [1.32 to 3.67] | 0.15 [-0.94 to 1.24] | 2.45 [1.28 to 3.62]
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Ponsegromab 100 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0090, MMRM analysis; 1-sided; Difference in LS Mean = 2.35, 90% CI 2-sided [0.72 to 3.97]
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: Ponsegromab 200 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.4987, MMRM analysis; 1-sided; Difference in LS Mean = 0, 90% CI 2-sided [-1.55 to 1.56]
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: Ponsegromab 400 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0100, MMRM analysis; 1-sided; Difference in LS Mean = 2.3, 90% CI 2-sided [0.68 to 3.92]

8. Secondary Outcome: Part A: Change From Baseline in Cancer-Related Cachexia Symptom Diary (CRCSD) Scores at Week 12: Appetite, Nausea and Physical Fatigue
Description: The CRCSD is a daily, self-reported questionnaire that measured severity of symptoms related to cancer cachexia: appetite, nausea, vomiting, and fatigue. Participants rated appetite, nausea and physical fatigue symptom every day, and weekly averages were calculated over the 7 days prior, from 0 to 10, where 0 = no symptom and 10 = worst possible symptom. Higher scores indicated more severe disease. CRCSD was analyzed using an MMRM model.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Part A: Placebo | Part A: Ponsegromab 100 mg | Part A: Ponsegromab 200 mg | Part A: Ponsegromab 400 mg
Number analyzed (Participants) | 24 | 30 | 26 | 27
Units on a scale
  Appetite | -0.23 [-0.83 to 0.37] | 0.20 [-0.36 to 0.76] | 0.23 [-0.37 to 0.82] | 0.69 [0.11 to 1.27]
  Nausea | -0.33 [-0.82 to 0.17] | 0.14 [-0.32 to 0.61] | 0.06 [-0.43 to 0.55] | -0.50 [-0.98 to -0.02]
  Physical Fatigue | -0.27 [-0.85 to 0.32] | 0.39 [-0.16 to 0.94] | 0.38 [-0.21 to 0.96] | -0.06 [-0.63 to 0.51]
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Ponsegromab 100 mg; Appetite: MMRM model included participant as a random term, and baseline, time (as a factor), baseline-by-time interaction, treatment and treatment-by-time interaction, type of therapy [platinum or not at randomization +/- 28 days], and type of cancer as fixed terms, with an unstructured covariance matrix and Kenwood-Roger degrees of freedom; Test type: Superiority; p = 0.1912, MMRM analysis; 1-sided; Difference in LS Mean = 0.43, 90% CI 2-sided [-0.38 to 1.24]
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: Ponsegromab 200 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.1866, MMRM analysis; 1-sided; Difference in LS Mean = 0.46, 90% CI 2-sided [-0.39 to 1.30]
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: Ponsegromab 400 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0349, MMRM analysis; 1-sided; Difference in LS Mean = 0.92, 90% CI 2-sided [0.09 to 1.75]
Statistical Analysis 4: Comparison: Part A: Placebo vs Part A: Ponsegromab 100 mg; Nausea: MMRM model included participant as a random term, and baseline, time (as a factor), baseline-by-time interaction, treatment and treatment-by-time interaction, type of therapy [platinum or not at randomization +/- 28 days], and type of cancer as fixed terms, with an unstructured covariance matrix and Kenwood-Roger degrees of freedom; Test type: Superiority; p = 0.8754, MMRM analysis; 1-sided; Difference in LS Mean = 0.47, 90% CI 2-sided [-0.20 to 1.14]
Statistical Analysis 5: Comparison: Part A: Placebo vs Part A: Ponsegromab 200 mg; [analysis description as in outcome 8, analysis 4]; Test type: Superiority; p = 0.8205, MMRM analysis; 1-sided; Difference in LS Mean = 0.38, 90% CI 2-sided [-0.31 to 1.08]
Statistical Analysis 6: Comparison: Part A: Placebo vs Part A: Ponsegromab 400 mg; [analysis description as in outcome 8, analysis 4]; Test type: Superiority; p = 0.3375, MMRM analysis; 1-sided; Difference in LS Mean = -0.17, 90% CI 2-sided [-0.86 to 0.51]
Statistical Analysis 7: Comparison: Part A: Placebo vs Part A: Ponsegromab 100 mg; Physical Fatigue: MMRM model included participant as a random term, and baseline, time (as a factor), baseline-by-time interaction, treatment and treatment-by-time interaction, type of therapy [platinum or not at randomization +/- 28 days], and type of cancer as fixed terms, with an unstructured covariance matrix and Kenwood-Roger degrees of freedom; Test type: Superiority; p = 0.9138, MMRM analysis; 1-sided; Difference in LS Mean = 0.66, 90% CI 2-sided [-0.14 to 1.45]
Statistical Analysis 8: Comparison: Part A: Placebo vs Part A: Ponsegromab 200 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority; p = 0.9011, MMRM analysis; 1-sided; Difference in LS Mean = 0.64, 90% CI 2-sided [-0.18 to 1.46]
Statistical Analysis 9: Comparison: Part A: Placebo vs Part A: Ponsegromab 400 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority; p = 0.6618, MMRM analysis; 1-sided; Difference in LS Mean = 0.21, 90% CI 2-sided [-0.61 to 1.02]

9. Secondary Outcome: Part A: Median Change From Baseline in CRCSD Scores at Week 12: Vomiting Frequency
Description: The CRCSD is a daily, self-reported questionnaire that measured severity of symptoms related to cancer cachexia: vomiting frequency. Participants rated vomiting frequency over the past 24 hours, from 0 to 30, where 0 = no symptom and 30 = worst possible symptom. Higher scores indicated more severe disease.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Part A: Placebo | Part A: Ponsegromab 100 mg | Part A: Ponsegromab 200 mg | Part A: Ponsegromab 400 mg
Number analyzed (Participants) | 24 | 30 | 26 | 27
Units on a scale | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0]

10. Secondary Outcome: Part A: Number of Participants With Treatment Emergent Adverse Events (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered a pharmaceutical product during the course of a clinical investigation. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product, whether or not thought to be related to the investigational product. TEAE were defined as any event that was not present before exposure to study drug, or any event already present that worsened in either intensity or frequency after exposure to study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included serious AEs and all non-SAEs.
Time Frame: From start of study drug on Day 1 maximum up to 4 weeks post last dose on Week 12 (maximum up to approximately Week 16)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Ponsegromab 100 mg | Part A: Ponsegromab 200 mg | Part A: Ponsegromab 400 mg
Number analyzed (Participants) | 45 | 46 | 46 | 50
Participants | 36 | 32 | 31 | 37

11. Secondary Outcome: Part A: Number of Participants With Incidence of Laboratory Test Abnormalities
Description: Laboratory test abnormality parameters included: hematology- hemoglobin (gram per deciliter [g/dL]), hematocrit (%), erythrocytes (10^12/Liter [L]) less than (<) 0.8*lower limit of normal (LLN); platelets (10^9/L) <0.5*LLN to more than (>) 1.75*upper limit of normal (ULN); leukocytes (10^9/L) <0.6*LLN to >1.5*ULN; lymphocytes, neutrophils (10^9/L) <0.8*LLN to >1.2*ULN. Clinical chemistry- bilirubin, glucose (mg/dL) >1.5*ULN; aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase (Units/L [U/L]) >3.0*ULN; protein, albumin (gram [g]/dL) <0.8*LLN; urea (mmol/L) >1.3xULN; creatinine (mg/dL) >1.3*ULN; sodium (milliequivalents [mEq]/L) <0.95*LLN; potassium (mEq/L) <0.9*LLN to >1.1*ULN.
Time Frame: Day 1 up to Week 12
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Ponsegromab 100 mg | Part A: Ponsegromab 200 mg | Part A: Ponsegromab 400 mg
Number analyzed (Participants) | 37 | 35 | 40 | 41
Participants | 26 | 24 | 29 | 28

12. Secondary Outcome: Part A: Number of Participants With Post-Baseline Vital Signs Meeting the Predefined Criteria
Description: Vital signs criteria included: supine systolic blood pressure (SBP) <90 millimeters of mercury (mmHg), increase and decrease in change of more than or equal to (>=) 30mmHg; supine diastolic blood pressure (DBP) <50 mmHg, increase and decrease in change of >= 20mmHg; pulse rate <40 beats per minute (bpm) to >120 bpm. Only rows which included at least 1 participant in any reporting group with abnormality were reported in this outcome measure.
Time Frame: Day 1 up to Week 12
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Ponsegromab 100 mg | Part A: Ponsegromab 200 mg | Part A: Ponsegromab 400 mg
Number analyzed (Participants) | 40 | 40 | 44 | 44
Participants
  Supine SBP Value < 90mmHg | 0 | 3 | 0 | 0
  Supine SBP Increase Change >= 30mmHg | 4 | 5 | 8 | 2
  Supine SBP Decrease Change >= 30mmHg | 2 | 6 | 5 | 4
  Supine DBP Value < 50mmHg | 0 | 1 | 0 | 0
  Supine SBP Increase Change >= 20mmHg | 4 | 4 | 3 | 4
  Supine DBP Decrease Change >= 20mmHg | 3 | 4 | 4 | 3
  Supine Pulse Rate Value > 120mmHg | 0 | 1 | 3 | 1

13. Secondary Outcome: Part A: Number of Participants With Clinically Significant Echocardiogram (ECG) Abnormalities
Description: ECG parameters included heart rate (HR), PR interval, QT interval, QTc corrected using Fridericia's formula (QTcF) and QRS complex. HR: RR (interval between 2 successive R waves on ECG) decrease >25% and to a VR (interval between QRS wave and T wave on ECG) >100, RR increase >25% and to a VR <50; PR interval: baseline less than or equal to (<=) 200 and % change >= 50%; QT interval: >450, >480, >500, increase from baseline >30, increase from baseline >60; QTcF: 470 < value <= 480, 480 < value <= 500, value > 500, 30 < change <= 60 and change >60; QRS complex: value >= 140, % change >=50%. Clinically significant values were determined by the investigator.
Time Frame: Day 1 up to Week 12
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Ponsegromab 100 mg | Part A: Ponsegromab 200 mg | Part A: Ponsegromab 400 mg
Number analyzed (Participants) | 45 | 46 | 46 | 50
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Part A: From start of study drug on Day 1 maximum up to 4 weeks post last dose on Week 12 (maximum up to approximately Week 16)
Description: Same event may appear as AE and SAE. What is presented are distinct events. Event may be categorized serious in 1 participant and non-serious in another, or participant may have experienced serious and non-serious event. Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. At this milestone (primary completion date) Part A safety analysis was final. Part B safety data will be reported at study completion date.
Groups:
- Part A: Placebo: Participants were randomized to receive placebo matching to Ponsegromab SC Q4W up to 12 weeks (total of 3 doses).
- Part A: Ponsegromab 100 mg: Participants were randomized to receive Ponsegromab 100 mg SC Q4W up to 12 weeks (total of 3 doses).
- Part A: Ponsegromab 200 mg: Participants were randomized to receive Ponsegromab 200 mg SC Q4W up to 12 weeks (total of 3 doses).
- Part A: Ponsegromab 400 mg: Participants were randomized to receive Ponsegromab 400 mg SC Q4W up to 12 weeks (total of 3 doses).
Arm/Group | Part A: Placebo | Part A: Ponsegromab 100 mg | Part A: Ponsegromab 200 mg | Part A: Ponsegromab 400 mg
All-Cause Mortality (participants affected / at risk) | 5/45 | 6/46 | 6/46 | 9/50
Serious Adverse Events (participants affected / at risk) | 11/45 | 15/46 | 10/46 | 20/50
Other Adverse Events (participants affected / at risk) | 25/45 | 19/46 | 19/46 | 24/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=45) | Part A: Ponsegromab 100 mg (N=46) | Part A: Ponsegromab 200 mg (N=46) | Part A: Ponsegromab 400 mg (N=50)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 2
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 1
Intestinal fistula infection (Infections and infestations) | 0 | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Pelvic abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 2 | 3
Pneumonia aspiration (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Anastomotic complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 3 | 3
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 2 | 2
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebral amyloid angiopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Diplegia (Nervous system disorders) | 0 | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Paraplegia (Nervous system disorders) | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=45) | Part A: Ponsegromab 100 mg (N=46) | Part A: Ponsegromab 200 mg (N=46) | Part A: Ponsegromab 400 mg (N=50)
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | 4 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 1 | 3
Constipation (Gastrointestinal disorders) | 4 | 3 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 8 | 3 | 4 | 5
Nausea (Gastrointestinal disorders) | 7 | 1 | 1 | 4
Vomiting (Gastrointestinal disorders) | 5 | 2 | 2 | 1
Asthenia (General disorders) | 1 | 1 | 3 | 4
Fatigue (General disorders) | 2 | 1 | 1 | 4
Oedema peripheral (General disorders) | 1 | 1 | 0 | 4
Pyrexia (General disorders) | 3 | 0 | 5 | 4
Pneumonia (Infections and infestations) | 3 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 3
Alanine aminotransferase increased (Investigations) | 3 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 4 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 6 | 0 | 6
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT05546476/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-07): https://cdn.clinicaltrials.gov/large-docs/76/NCT05546476/SAP_001.pdf